CLINICAL TRIAL: NCT04738097
Title: Ticagrelor Plus Aspirin vs Clopidogrel Plus Aspirin in Mild Non-cardioembolic Ischemic Stroke: A Randomized, Active Comparator Arm, Outcome Assessor Blind, Controlled, Feasibility Study
Brief Title: Efficacy of Ticagrelor Plus Aspirin in Mild Non-cardioembolic Ischemic Stroke
Acronym: TACAMINIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Athena Sharifi Razavi, Assistant professor in Neurology, Mazandaran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4164
Record Dates: First submitted 2021-01-31; First posted 2021-02-04 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack
Keywords: minor stroke; secondary prevention; ticagrelor; aspirin; recurrence; non-cardioembolic; antiplatelet
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient; Recurrence | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Experimental): Intervention group will be treat with ASA 325 mg stat and ticagrelor 180 mg stat, then ASA 80 mg daily and ticagrelor 90 mg BID for 21 days.
  Interventions: Drug: Ticagrelor 90mg
- control (Active Comparator): control group will be treat with ASA 325 mg stat and clopidogrel 300 mg stat, then ASA 80 mg and clopidogrel 75 mg daily for 21 days.
  Interventions: Drug: Clopidogrel 75 mg

INTERVENTIONS:
Drug: Ticagrelor 90mg — ASA 325 mg stat and ticagrelor 180 mg stat, then ASA 80 mg daily and ticagrelor 90 mg BID for 21 days.Treatment will be continue with ASA 80 until 3 months.
  Other Names: Ticer
  Arms: intervention
Drug: Clopidogrel 75 mg — ASA 325 mg stat and clopidogrel 300 mg stat, then ASA 80 mg and clopidogrel 75 mg daily for 21 days.Treatment will be continue with ASA 80 until 3 months.
  Other Names: Osvix
  Arms: control

SUMMARY:
This is a randomized, controlled, active comparator arm, outcome assessor blind, parallel group design on 90 patient with diagnosis of ischemic stroke admitted in Bou-Ali Sina Hospital, Sari,Iran.The aim of study is assess the efficacy of ticagrelor plus aspirin in reduce of minor non-cardioembolic ischemic stroke or high risk TIA recurrence during first 3 months.

DETAILED DESCRIPTION:
This is a randomized, controlled, parallel, active comparator arm, outcome assessor blind, feasibility study. The aim of study is assess the efficacy of ticagrelor plus aspirin in reduce of minor non-cardioembolic ischemic stroke or high risk TIA recurrence during first 3 months after primary event. 90 patient with diagnosis of ischemic stroke admitted in Bou-Ali Sina Hospital, Sari, Iran will be randomized to intervention or control group by using 4 block randomization method. Inclusion criteria is : age>40, signing inform consent, recent ischemic stroke within 24 h, diagnosed by brain CT or MRI mild stroke with NIHSS =<8 and no evidence of large infarct in brain imaging.,high risk TIA with ABCD >4, no cardioembolic source such as low E/F, MS, AF ,... no specific etiology such as dissection, vasculitis, ... no carotid stenosis > 50 % in side of involvement. Exclusion criteria is :history of hypersensitivity to consumptive drug any indication for anticoagulant therapy acute phase treatment with intravenous thrombolysis or thrombectomy any contraindication for consumptive drug history of intracranial hemorrhage history of GI bleeding during past 6 m candidate for endarterectomy history of coagulopathy active hemorrhagic diathesis during randomization. Patients in control group will be treat with standard minor ischemic stroke regiment including ASA 325 mg stat and clopidogrel 300 mg stat, then ASA 80 mg and clopidogrel 75 mg daily for 21 days. Intervention group will be treat with ASA 325 mg stat and ticagrelor 180 mg stat, then ASA 80 mg daily and ticagrelor 90 mg BID for 21 days. Then all groups will be treat with ASA 80 mg daily after day 21. Three fallow up visit plan by a neurologist or neurology resident on month 1 and 3.Clinical data including NIHSS score, MRS score and other data will record on case report form. Stroke recurrence or cardiovsacular event is efficacy end point. Major bleeding according to STIH criteria is study safety end point. Primary outcome is ischemic stroke recurrence during first 3 months after first event documented by new lesion on brain CT or MRI. Secondary outcome is major hemorrhagic events, stroke recurrence during first 30 days and any cardiovascular event during first 3 month.

ELIGIBILITY:
Inclusion Criteria:

* signing inform consent,
* recent ischemic stroke within 24 h,
* diagnosed by brain CT or MRI mild stroke with NIHSS =<8 and no evidence of large infarct in brain imaging
* high risk TIA with ABCD >4,
* no cardioembolic source such as low E/F, MS, AF ,...
* no specific etiology such as dissection, vasculitis, ...
* no carotid stenosis > 50 % in side of involvement

Exclusion Criteria:

* history of hypersensitivity to consumptive drug
* any indication for anticoagulant therapy
* acute phase treatment with intravenous thrombolysis or thrombectomy
* any contraindication for consumptive drug
* history of intracranial hemorrhage
* history of GI bleeding during past 6 m
* candidate for endarterectomy
* history of coagulopathy
* active hemorrhagic diathesis during randomization

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-08-08 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
ischemic stroke recurrence | first 3 months after first event
  recording new event based on new lesion on brain CT scan or MRI

SECONDARY OUTCOMES:
Major hemorrhagic event | during first 30 days
  Major bleeds were defined according to the International Society of Thrombosis and Hemostasis (ISTH)
ischemic stroke recurrence | first 1 month after first event
  recording new event based on new lesion on brain CT scan or MRI
cardiovascular events | during first 3 months after first event
  any proven cardiovascular event

CONTACTS AND LOCATIONS:
Overall Officials: Athena Sharifi-Razavi, Principal Investigator — Mazandaran University of Medical science
Locations (2):
- Iran (2):
  - Athena Sharifi Razavi, Sari, Mazandaran
  - Bou-Ali Sina hospital , Mazandarn University of Medical Science, Sari

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared by request to principal investigator for scientifical reseasons
Supporting Information: SAP, ICF
Time Frame: 6 months after publishing study results
Access Criteria: requested by a scientifically person, who plan for similar protocol study

REFERENCES:
- See also: published study protocol article — https://www.neurology-asia.org/articles/neuroasia-2023-28(3)-535.pdf